CLINICAL TRIAL: NCT00547274
Title: Dyslipidemia in Type 2 Diabetes (0767-034)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0767-034; 2007_635; MK-0767-034
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type II; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — MK0767

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0767

SUMMARY:
The purpose of the study is to compare the lipid-altering effects of MK0767, glipizide, and pioglitazone after 12 weeks of treatment.

This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant females
* Age greater than or equal to 21 years
* Stop current diabetes therapy (if applicable)
* Stop current statin therapy (if applicable)

Exclusion Criteria:

* History of type 1 diabetes mellitus or ketoacidosis who are currently being treated with insulin
* Patients on a weight loss program with ongoing weight loss, or starting an intensive exercise program within the last four weeks
* Patients requiring treatment with corticosteroids for more than 14 consecutive days
* Patients taking warfarin or warfarin-like anti-coagulants
* Patients undergoing surgery within 30 days of Visit 1
* Patients with Hepatitis B, Hepatitis C, active liver or gallbladder disease
* Patients with history of pancreatitis or uncontrolled high blood pressure

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2003-07; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC